CLINICAL TRIAL: NCT00916032
Title: Pharmacokinetic Comparison of 3000 IU Advate (rAHF-PFM) (Using One 3000 IU Potency Vial) With 3000 IU Advate (rAHF PFM) (Using Two 1500 IU Potency Vials) in Previously Treated Patients With Severe Hemophilia A: a Phase 4, Open-label, Prospective, Randomized, Controlled, Crossover, Multiple Center Study
Brief Title: Pharmacokinetic Study of ADVATE 3000 IU in Previously Treated Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060801; 2008-007347-13 (EudraCT Number)
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): One infusion using a 3000 IU potency vial of Advate dissolved and administered in 5 mL diluent followed by a second infusion of two 1500 IU potency vials of Advate dissolved in 5 mL diluent each (administered in 10 mL diluent in total)
  Interventions: Biological: Octocog alfa (recombinant human coagulation factor VIII) [ADVATE]
- 2 (Active Comparator): One infusion of two 1500 IU potency vials of Advate dissolved in 5 mL diluent each (administered in 10 mL diluent in total) followed by a second infusion of one 3000 IU potency vial of Advate dissolved and administered in 5 mL diluent
  Interventions: Biological: Octocog alfa (recombinant human coagulation factor VIII) [ADVATE]

INTERVENTIONS:
Biological: Octocog alfa (recombinant human coagulation factor VIII) [ADVATE] — Participants will receive 3000 IU Advate using one 3000 IU potency vial dissolved in 5 mL diluent followed by two 1500 IU potency vials dissolved in 5 mL diluent each (administered in 10 mL diluent in total) or the alternate sequence
  Other Names: ADVATE; Antihemophilic Factor (Recombinant)- Plasma/albumin free method (rAHF-PFM)

SUMMARY:
The objective of this clinical study is to compare the pharmacokinetic parameters of 3000 IU Advate using one 3000 IU potency vial dissolved in 5 mL diluent with that of 3000 IU Advate using two vials of 1500 IU potency dissolved in 5 mL diluent each (administered in 10 mL diluent in total) in previously treated patients with severe hemophilia A (factor VIII level < 1%).

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 to 65 years old, at the time of screening
* Participant has provided signed informed consent
* Participant has severe hemophilia A, defined by a baseline FVIII level < 1% of normal, as tested at screening at the central laboratory
* Participant's weight is between 55-65 kg
* Participant was previously treated with FVIII concentrate(s) for a minimum of 150 exposure days prior to study entry
* If Participant is HIV positive, he must be immunocompetent as determined with a CD4 count ≥ 200 cells/mm³ (CD4 count at screening)
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Participant has a detectable FVIII inhibitor at screening, with a titer ≥ 0.4 Bethesda unit (BU) (Nijmegen modification of the Bethesda Assay) measured at the central laboratory
* Participant has a history of FVIII inhibitors with a titer ≥ 0.4 BU (by Nijmegen assay) or ≥ 0.5 BU (by Bethesda Assay) at any time prior to screening
* Participant has undergone a surgery within 21 days prior to screening or within 6 weeks prior to the anticipated first pharmacokinetics(PK) infusion
* Participant has an abnormal renal function (serum creatinine > 1.5 mg/dL)
* Participant has active hepatic disease (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >5 times the upper limit of normal)
* Participant has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) > 1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly, and history of esophageal varices
* Participant has clinical and/or laboratory evidence of abnormal hemostasis from causes other than hemophilia A (eg, late-stage chronic liver disease, immune thrombocytopenia purpura)
* Participant is currently receiving, or is scheduled to receive during the course of the clinical study, an immunomodulating drug other than anti-retroviral chemotherapy (eg, alfa-interferon, or corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day)
* Participant has a known hypersensitivity to mouse or hamster proteins
* Participant has participated in another clinical study involving an investigational product or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product or investigational device during the course of this clinical study
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures
* Participant is a member of the team conducting this clinical study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, or parents) as well as employees of the investigator or site personnel conducting the clinical study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Sofia, Bulgaria
- Russia (3):
  - Kirov
  - Moscow
  - Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted in Russia and Bulgaria at 4 clinical sites.
Pre-assignment Details: 29 participants were enrolled. Six participants discontinued, (four were screen failures and two were withdrawn before randomization). Therefore 23 participants were randomized.
Groups:
- Two 1500 IU Vials Then One 3000 IU Vial: Participants received via intravenous (IV) infusion 3000 International Units (IU) Advate using two 1500 IU potency vials dissolved in 5 mL diluent each (administered in 10 mL diluent in total) followed by one 3000 IU potency vial dissolved in 5 mL diluent.
- One 3000 IU Vial Then Two 1500 IU Vials: Participants received via intravenous (IV) infusion 3000 International Units (IU) Advate using one 3000 IU potency vial dissolved in 5 mL diluent followed by two 1500 IU potency vials dissolved in 5 mL diluent each (administered in 10 mL diluent in total)
Period: Overall Study
Arm/Group | Two 1500 IU Vials Then One 3000 IU Vial | One 3000 IU Vial Then Two 1500 IU Vials
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive via intravenous infusion 3000 International Units (IU) Advate using either one 3000 IU potency vial dissolved in 5 mL diluent followed by two 1500 IU potency vials dissolved in 5 mL diluent each (administered in 10 mL diluent in total) or the alternate sequence.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 14
  Russian Federation | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to 48 Hours (AUC 0-48h). Chromogenic Assay
Description: Computed using the linear trapezoidal method.
Time Frame: Within 30 minutes prior to the start of the infusion; and after the end of the infusion at 15, 30 minutes, and 1, 3, 6, 9, 24, 28, 32, and 48 hours.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU·h)/dL
Groups:
- One 3000 International Unit (IU) Vial: Participants received via intravenous (IV) infusion 3000 International Units (IU) Advate using one 3000 IU potency vial dissolved in 5 mL diluent
- Two 1500 IU Vials: Participants received via intravenous (IV) infusion 3000 International Units (IU) Advate using two 1500 IU potency vials dissolved in 5 mL diluent each (administered in 10 mL diluent in total)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU·h)/dL | 1158 (335) | 1264 (364)
Statistical Analysis 1: Comparison: One 3000 International Unit (IU) Vial vs Two 1500 IU Vials; Test type: Superiority or Other; p = 0.103, paired t-test done on the Log(AUC 0-48h)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to 48 Hours (AUC 0-48h). One-stage Activated Partial Thromboplastin Time (aPTT) Assay
Description: Computed using the linear trapezoidal method.
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU·h)/dL
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU·h)/dL | 1129 (310) | 1226 (358)
Statistical Analysis 1: Comparison: One 3000 International Unit (IU) Vial vs Two 1500 IU Vials; Test type: Superiority or Other; p = 0.162, paired t-test done on the Log(AUC 0-48h)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to Infinity (AUC 0-infinity). Chromogenic Assay
Description: The total area under the plasma concentration versus time curve when the concentration is extrapolated to zero using the slope of the β-phase of the model.
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU·h)/dL
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU·h)/dL | 1267 (395) | 1383 (437)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to Infinity (AUC 0-infinity). One-stage aPTT Assay
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU·h)/dL
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU·h)/dL | 1235 (364) | 1348 (427)

5. Secondary Outcome: Incremental Recovery at Cmax - Chromogenic Assay
Description: Determined as the highest Factor VIII (FVIII) activity achieved post-infusion
Time Frame: Within 30 minutes prior to the start of the infusion; and after the end of the infusion at 15, 30 minutes, and 1, 3 hours.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU/dL)/(IU/kg) | 1.81 (0.40) | 2.04 (0.34)

6. Secondary Outcome: Incremental Recovery at Cmax - One-stage aPTT Assay
Description: Determined as the highest FVIII activity achieved post-infusion
Time Frame: as for outcome 5
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU/dL)/(IU/kg) | 1.75 (0.43) | 1.96 (0.32)

7. Secondary Outcome: Incremental Recovery at 30 Minutes- Chromogenic Assay
Description: Change in factor VIII concentration from pre-infusion to 30 minutes post-infusion
Time Frame: 30 minutes pre-infusion and 30 minutes post-infusion
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU/dL)/(IU/kg) | 1.62 (0.42) | 1.84 (0.40)

8. Secondary Outcome: Incremental Recovery at 30 Minutes- One-stage aPTT Assay
Description: Change in factor VIII concentration from pre-infusion to 30 minutes post-infusion
Time Frame: 30 minutes pre-infusion and 30 minutes post-infusion
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
(IU/dL)/(IU/kg) | 1.64 (0.43) | 1.90 (0.32)

9. Secondary Outcome: Elimination Phase Half-life- Chromogenic Assay
Description: calculated as log_e2/λ, where λ is the regression slope in the terminal phase of the least absolute deviations regression model
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
hour | 13.27 (4.05) | 12.84 (4.31)

10. Secondary Outcome: Elimination Phase Half-life- One-stage aPTT Assay
Description: as for outcome 9
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
hour | 13.80 (3.95) | 13.50 (2.81)

11. Secondary Outcome: FVIII Clearance- Chromogenic Assay
Description: computed as the dose divided by total AUC
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mL/(kg·h)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
mL/(kg·h) | 4.57 (1.75) | 3.99 (1.53)

12. Secondary Outcome: FVIII Clearance- One-stage aPTT Assay
Description: Computed as the dose divided by total AUC
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mL/(kg·h)
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
mL/(kg·h) | 4.66 (1.81) | 4.06 (1.46)

13. Secondary Outcome: Mean Residence Time (MRT)- Chromogenic Assay
Description: Computed as total area under the first moment curve (Total AUMC) divided by the total area under the concentration versus time curve (Total AUC)
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
hour | 17.02 (5.37) | 16.84 (5.81)

14. Secondary Outcome: Mean Residence Time (MRT)- One-stage aPTT Assay
Description: as for outcome 13
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
hour | 16.95 (4.77) | 17.16 (4.65)

15. Secondary Outcome: Volume of Distribution at Steady State- Chromogenic Assay
Description: computed as Clearance (CL) * Mean residence time (MRT)
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
dL/kg | 0.72 (0.23) | 0.61 (0.13)

16. Secondary Outcome: Volume of Distribution at Steady State- One-stage aPTT Assay
Description: computed as CL * MRT
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
dL/kg | 0.74 (0.19) | 0.64 (0.11)

17. Secondary Outcome: Factor VIII (FVIII) Maximum Plasma Concentration (C-max)- Chromogenic Assay
Description: Determined as the highest FVIII activity achieved post-infusion.
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
IU/dL | 94 (21) | 101 (18)

18. Secondary Outcome: Factor VIII (FVIII) Maximum Plasma Concentration (C-max)- One-stage aPTT Assay
Description: Determined as the highest FVIII activity achieved post-infusion.
Time Frame: as for outcome 1
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Number analyzed (Participants) | 23 | 23
IU/dL | 91 (21) | 98 (20)

ADVERSE EVENTS:
Time Frame: Throughout the study period, approximately 10 months
Arm/Group | One 3000 International Unit (IU) Vial | Two 1500 IU Vials
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication of the main/primary endpoint or ≤24 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) prior to submission for publication, and shall review and if necessary amend the manuscript in ≤30 days